CLINICAL TRIAL: NCT04990921
Title: A Phase 2 Study of Palliative Radiation in Combination with Pembrolizumab in Subjects with Unresectable Metastatic Stage IV Breast Cancer: Twisted Pink
Brief Title: Study of Palliative Radiation Combined with Pembrolizumab in Unresectable Metastatic Stage IV Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Riley, Principal Investigator, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Twisted Pink Foundation
Record Dates: First submitted 2021-06-23; First posted 2021-08-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The primary objective is to evaluate the efficacy of SBRT in combination with pembrolizumab as assessed by Overall Response Rate in subjects with stage IV breast cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Palliative Radiation in Combination with Pembrolizumab (Experimental): Stereotactic radiation therapy will be delivered using either linac-based SBRT using 10x flattening filter-free (FFF) photons or Cyberknife Pencil Beam Technology utilizing 6X photons. Treatment will be delivered in 1-5 fractions. Fractionation and total dose (1500 - 3000 cGy) will depend on the site of disease, previous radiation treatment, and patient symptomatology.
  Pembrolizumab is supplied as pembrolizumab 100 mg/4 mL vials (25 mg/mL) solution for intravenous infusion. Pembrolizumab at a dose of 200 mg will be administered intravenously every 3 weeks (± 3 days).
  Interventions: Combination Product: Palliative Radiation and Pembrolizumab

INTERVENTIONS:
Combination Product: Palliative Radiation and Pembrolizumab — Stereotactic radiation therapy will be administered as clinically indicated.
  Other Names: Keytruda

SUMMARY:
This is a phase 2, open-label, single-arm trial designed to evaluate the efficacy and safety of stereotactic body radiation therapy (SBRT) in combination with pembrolizumab following disease progression after two prior lines of standard therapy in unresectable metastatic stage IV breast cancer

DETAILED DESCRIPTION:
This study will enroll subjects who are female aged > 18 years at the time of informed consent with histologically confirmed diagnosis of breast cancer (unresectable or metastatic stage IV breast cancer). Subjects must have measurable disease and be a candidate for palliative stereotactic body radiation therapy (SBRT). Subjects must have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0, 1, or 2 and adequate hematologic, hepatic, renal, and coagulation function. Subject must also have received two prior lines of FDA-approved therapy. Triple negative patients must have had prior exposure to taxane therapy either in the neoadjuvant/adjuvant or metastatic setting. ER + positive patients must have had prior cyclin dependent kinase (CDK) 4/6 inhibitor therapy. Her2 overexpressed patients must have had prior therapy with trastuzumab and ado-trastuzumab (TDM-1).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject has provided informed consent/assent prior to initiation of any study specific activities/procedures.

  2. Female age ≥ 18 years at the time of informed consent. 3. Histologically confirmed diagnosis of breast cancer. 4. Disease stage: unresectable or metastatic stage IV breast cancer. 5. Candidate for palliative SBRT independent from study enrollment 6. Measurable disease, defined as at least 1 visceral or nodal/soft tissue breast cancer lesion that can be accurately and serially measured in at least 1 dimension and for which the longest diameter is ≥ 10 mm as measured by Computer Tomography scan or Magnetic Resonance Imaging. Lymph nodes must measure ≥ 15 mm in their short axis to be considered measurable by Computer Tomography scan or Magnetic Resonance Imaging or Positron Emission Tomography-CT.

  7. If subject received major surgery, must have recovered adequately from toxicity and/or complications from the intervention prior to enrollment.

  8. Subject must have received two prior lines of therapy and include a taxane in the adjuvant/neoadjuvant or metastatic setting.
  1. Triple negative breast cancer patients must have received two lines of chemotherapy in the metastatic setting.
  2. ER+/ PR+, ER-/PR+, and ER+/PR- must have received prior Cyclin Dependent Kinase 4/6 Inhibitor in combination with Aromatase Inhibitor or fulvestrant. However, ER+/Her2 overexpressed patients are not required to have received CDK 4/6 inhibitor.
  3. Her2 overexpressed breast cancer must have had prior trastuzumab/per (in the neoadjuvant/adjuvant or metastatic setting, and prior Ado-trastuzumab TDM1 therapy.

     9. Adequate organ function determined within 14 days prior to enrollment, defined as follows:
     * Absolute neutrophil (ANC) >1.5 x 109/L
     * Platelet count>50 x 109/L
     * Hemoglobin>8 g/dL
     * Serum creatinine <2.0 x upper limit of normal
     * Serum bilirubin < 2.0 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 2.0 x ULN
     * Aspartate aminotransferase (AST) <2.5 x ULN OR <5 x ULN for subject with liver metastases
     * Alanine aminotransferase (ALT) <2.5 x ULN OR <5 x ULN for subject with liver metastases
     * International normalization ratio (INR) or prothrombin time (PT) <1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and partial thromboplastin time (PTT)/activated PTT (aPTT) is within therapeutic range of intended use of anticoagulants
     * Lactate dehydrogenase (LDH) levels ≤ 1.5 X upper limit of normal (ULN) within 28 days prior to enrollment
     * Female subject of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If the urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
     * ECOG performance status of 0, 1 or 2.

     Exclusion Criteria:

  <!-- -->

  1. > 4 Clinically active cerebral metastases. Subjects cerebral metastases may be enrolled, provided that there are less than 4 lesions as these may serve as a site of pallative SBRT
  2. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
  3. Any active autoimmune disease that in the judgement of the PI or sub-I could be significantly worsened by pembrolizumab
  4. Evidence of clinically significant immunosuppression such as the following:

     * diagnosis of immunodeficiency;
     * concurrent opportunistic infection;
     * receiving systemic immunosuppressive therapy (> 2 weeks) or within 7 days prior to the first dose of study treatment, including oral steroid doses > 20 mg/day of prednisone or equivalent Subjects that require intermittent use of bronchodilators or local steroid injection will not be excluded from the study.
  5. Subject has known sensitivity to any of the products or components to be administered during dosing
  6. Known human immunodeficiency virus (HIV) disease.
  7. Known acute or chronic hepatitis B or hepatitis C infection.
  8. Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. Subjects who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of Graft versus Host Disease.
  9. Has a known history of active Bacillus tuberculosis.
  10. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
  11. Those patients who would not otherwise have an indication for palliative SBRT
  12. Prior therapy with tumor vaccine (unless administered in the adjuvant setting).
  13. Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study.
  14. Expected to require other cancer therapy while on study with the exception of local radiation treatment to the site of bone and other metastasis for palliative pain management. Concurrent endocrine therapy or trastuzumab therapy is allowed if clinically indicated. Concurrent bone modifying agents (including denosumab or zoledronic acid) is allowed for patients with bone metastases.
  15. Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment or 4 months after the last dose of pembrolizumab
  16. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment or 4 months after the last dose of pembrolizumab, whichever is later. Note: Women not of childbearing potential are defined as:

      * postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone follicule stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.); OR
      * have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening; OR
      * has a congenital or acquired condition that prevents childbearing.
  17. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2031-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 3.0 years
  Overall Response Rate (complete response [CR]+partial response [PR] by investigator assessment using modified RECIST v1.1) at week 24

SECONDARY OUTCOMES:
Secondary Outcome Measures-Best Overall Response Rate | 3.0 years
  Best Overall Response Rate (complete response [CR]+partial response [PR] by investigator assessment using modified RECIST v1.1)
Secondary Outcome Measures-Progression-free Survival | 3.0 years
  Progression-free Survival (PFS)
Secondary Outcome Measures-Incidence of treatment-emergent and treatment-related adverse events | 3.0 years
  Incidence of treatment-emergent and treatment-related adverse events as defined by

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Riley, MD, Principal Investigator — UL Health Brown Cancer Center Deputy Director, Health Affairs
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Data identifying the subjects and subject research records that are maintained in the Clinical Trials Office (CTO) will be made available to the study sponsor or its authorized representatives during monitoring visits. Many source documents may contain identifiable information.
  During internal audits, members of the James Graham Brown Cancer Center (JGBCC) Data Safety Monitoring Committee will have access to subject's research records maintained in the CTO. If required, these records will be made available to the FDA, Office for Human Research Protections (OHRP), Office of Civil Rights, and other authorized local/state/federal agencies.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available during the 3 year period of enrollment until long term analyses is complete and the study is terminated.